CLINICAL TRIAL: NCT07094932
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Trial in Healthy Adult Participants to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBD09 With an 84-day Period of Fixed Daily Dosing
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBD09
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gates Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gates MRI-TBD09-103
Record Dates: First submitted 2025-07-29; First posted 2025-07-31 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-10

CONDITIONS: Healthy Adult Participants
Keywords: Mycobacterium tuberculosis; TBD09; Fixed daily dosing; Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TBD09 (Active Comparator): Participants will be randomized to receive TBD09 once daily.
  Interventions: Drug: TBD09
- Placebo (Placebo Comparator): Participants will be randomized to receive placebo once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TBD09 — TBD09 will be administered orally
  Arms: TBD09
Drug: Placebo — Placebo will be administered orally
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multiple dose trial of TBD09, administered to healthy adult participants to assess safety, tolerability, and pharmacokinetics up to 84 days of fixed daily dosing of TBD09. The trial will be conducted with two cohorts, with participants enrolled in parallel and randomized to receive either TBD09 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Is healthy as determined by the Investigator via medical history and clinical examination before enrollment in the trial.
* Can understand and comply with the trial and site procedures, understand the risks involved in the trial, and provide written informed consent before the first trial-specific procedure
* Can complete all Screening period evaluations and stay in the clinical research facility for the duration of the inpatient periods of the trial.
* Has body mass index (BMI) between 18 and 32 kg/m^2 (kilograms per square meter), inclusive, and body weight not less than 50 kg at Screening.
* Has resting vital signs within the following ranges at Screening and Day -1:

  1. Systolic blood pressure (SBP) >= 100 mmHg (millimeters of mercury) and <= 140 mmHg
  2. Diastolic blood pressure (DBP) >= 60 mmHg and <= 90 mmHg
  3. Heart rate between 45 and 100 beats per minute (bpm)
* Has a 12-lead ECG consistent with normal cardiac conduction and function at Screening, including: HR between 45 and 100 bpm (inclusive); QTcF (QT Interval Corrected Using Fridericia's Formula) ≤450 ms (milliseconds) for males and ≤470 ms for females; QRS interval <120 ms; PR interval <220 ms; and morphology consistent with healthy cardiac conduction.
* Is a nonsmoker within the previous 90 days before Screening, with a negative urine cotinine test at the time of Screening, and does not use tobacco-containing, or nicotine-containing products, including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, e-cigarettes, nicotine patch, or nicotine gum.
* Has clinical chemistry (fasted for at least 8 hours), coagulation, and complete urinalysis results at Screening within the reference ranges for the testing laboratory unless the out-of-range results are deemed not clinically significant by the Investigator or designee, and documented as such in source documents.
* Has negative results for hepatitis B surface antigen (HBsAg) and hepatitis C virus antibody (HCV Ab) at Screening.
* Has negative test results for human immunodeficiency virus (HIV) antibody at Screening.
* Has a negative urine drug screen result at Screening and on Day -1.
* Has a negative urine alcohol screen result on Day -1.
* Has a hemoglobin A1c (HbA1c) result less than 5.7% at Screening.
* Has a thyroid stimulating hormone (TSH) level within the reference range for the testing laboratory at Screening.
* Has an absolute neutrophil count (ANC) greater than or equal to 2,000 neutrophils per microliter of blood.
* Has clinical hematology results for total white blood cell count, absolute lymphocyte count, hemoglobin, red blood cell count, and platelet count within the reference ranges for the testing laboratory at Screening.
* If individual's assigned sex at birth is female, they must have negative urine and serum pregnancy tests at Screening, and be of non-childbearing potential based on either of the following:

  1. Is post-menopausal defined as amenorrhea for at least 12 months in absence of any exogenous hormonal treatments and follicle stimulating hormone (FSH) levels in the laboratory-defined postmenopausal range, or,
  2. Reports being surgically sterilized (ie, tubal ligation, hysterectomy, bilateral oophorectomy/salpingectomy), and provides written documentation [(ie, medical record(s)], where feasible, to document such procedure(s) to the Principal Investigator. The site must make documented attempts to obtain medical records. If records cannot be retrieved, a participant may be enrolled at the Principal Investigator's discretion.
* If individual is assigned male sex at birth, is not sterilized, and is sexually active with a female partner of childbearing potential, agrees to use condoms from Day -1 through 90 days after the last dose of study drug. They must also agree to not donate sperm during the trial and for 3 months (90 days) after receiving the last dose of study drug.
* Agrees to follow lifestyle and dietary restrictions.

Exclusion Criteria:

* Has current or past history of a clinically significant cardiovascular, cerebrovascular, respiratory, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease, as determined by the Investigator.
* Has history of or Screening findings of peripheral neuropathy, such as numbness or abnormal reflexes.
* Has history of or Screening findings of abnormalities of vision, including corrected visual acuity worse than 20/25 in either eye based on Screening assessment using Snellen chart and Rosenbaum pocket chart, or color vision impairment based on Screening assessment using Ishihara plates. Candidates with ametropia corrected to 20/25 or better do not have to be excluded.
* Has history of or has clinically relevant cardiovascular disorder, such as heart failure, coronary artery disease, controlled or uncontrolled hypertension, arrhythmia, tachyarrhythmia, prolonged QT syndrome, or presence of symptom(s) strongly suggestive of such a problem, such as exertional chest pressure/pain or unexplained syncope.
* Had an active malignancy within 5 years from Screening, except basal cell or squamous cell skin cancers. Any history of breast cancer or melanoma will be exclusionary.
* Has history of any drug abuse within 1 year prior to Screening or has used any hard drugs (such as cocaine, phencyclidine [PCP], natural and synthetic opiates, and amphetamine derivatives) within 1 year prior to Screening. Individuals that have taken an opioid or amphetamine medication within the previous year prior to Screening that was prescribed by a healthcare provider will not be excluded unless they are currently taking the medication at the time of Screening.
* Had any surgical or medical condition or history that, in the opinion of the Investigator, may potentially alter the absorption, metabolism, or excretion of study treatment, such as, but not limited to, gastric bypass, sleeve, banding surgery, or gastric or duodenal ulcers
* Is taking any of the following prohibited medications or vaccinations:

  1. Any prescription or over-the-counter medication, vitamin or dietary supplement, or herbal product within 14 days prior to Day -1.
  2. Received any vaccination within 28 days prior to Day -1, including COVID-19 vaccination.
* Has a contraindication to study drugs or its excipients and/or history of a clinically significant allergic or anaphylactic reaction to any medication.
* Has participated in other trials involving administration of an investigational drug, vaccine or device within 30 days or 5 half-lives, whichever is longer, before Day -1 for the current trial and during participation in the current trial.
* Has a positive polymerase chain reaction (PCR) for COVID-19/SARS-CoV-2 on Day -1.
* Has a condition that the Investigator believes would interfere with the participant's ability to provide written informed consent, comply with trial instructions, or which might confound the interpretation of the trial results or put the participant at undue risk.
* Has donated blood within 2 months before Screening or planning to donate blood during the trial or within 12 weeks after the final visit.
* Has previously participated in a clinical trial involving TBD09.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-01-11 (Actual); Study Completion 2026-01-11 (Actual)

PRIMARY OUTCOMES:
Proportion of participants reporting treatment-emergent adverse events (TEAEs), serious AEs (SAEs), AEs of special interest (AESIs), and AEs leading to withdrawal of study drug after multiple administrations of TBD09. | Up to 92 days
Number of participants with clinically significant changes from baseline in safety laboratory measures | Day 1 through Day 92
Number of participants with clinically significant changes from baseline in vital signs | Day 1 through Day 92
Number of participants with clinically significant changes from baseline in electrocardiogram (ECG) parameters | Day 1 through Day 92

SECONDARY OUTCOMES:
Maximum plasma drug concentration (Cmax) of TBD09 in treated participants | Day 1
Time to maximal concentration (Tmax) of TBD09 in treated participants | Day 1
Area Under the concentration time curve from Zero to 24 hours (AUC 0-24) of TBD09 in treated participants | Day 1
Tmax of TBD09 in treated participants | Day 84
Cmax of TBD09 in treated participants | Day 84
Area Under the concentration time curve from the time of dosing to the time of the last measurable concentration (AUC last) of TBD09 in treated participants | Day 84
Minimum plasma drug concentration (Cmin) of TBD09 in treated participants | Day 84
Accumulation ratio (area under plasma concentration-time curve over dosing interval [AUCtau] / AUC0-24) of TBD09 in treated participants. Day 84 vs Day 1 | Day 84

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No